CLINICAL TRIAL: NCT05028127
Title: An Open-Label, Parallel-Group, Single-Dose Study to Evaluate the Relative Bioavailability and Tolerability of 160mg Subcutaneous Bimekizumab in Healthy Subjects
Brief Title: A Study to Evaluate the Relative Bioavailability and Tolerability of Bimekizumab in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Celltech (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UP0031
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08-01

CONDITIONS: Healthy Volunteers
Keywords: Bimekizumab; Phase 1
MeSH Terms: interventions — bimekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bimekizumab dosage regimen 1 (Experimental): Subjects participating in the study will be receiving assigned bimekizumab dosage regimen 1 during the Treatment Period.
  Interventions: Drug: Bimekizumab
- Bimekizumab dosage regimen 2 (Experimental): Subjects participating in the study will be receiving assigned bimekizumab dosage regimen 2 during the Treatment Period.
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Drug: Bimekizumab — Subjects will be receiving bimekizumab at pre-specified time-points.
  Other Names: UCB4940; BKZ

SUMMARY:
The purpose of the study to determine the relative bioavailability of bimekizumab in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female aged ≥18 years and ≤65 years at the Screening Visit
* Female subjects of child bearing potential must have a negative serum pregnancy test at the Screening Visit, which is confirmed to be negative by urine testing prior to the first dose of the Investigational Medicinal Product (IMP). Female subjects of childbearing potential must agree to use a highly effective method of birth control during the study and for a period of 20 weeks after their last dose of the IMP
* Subject must be in good health (physically and mentally) as determined by the Investigator on the basis of medical history (any chronic and acute illness), physical examination, vital signs, 12-lead ECG, and laboratory screening tests during the Screening Period
* Subject has a body weight of 45 to 90 kg (inclusive) and body mass index (BMI) between 19 and 28 kg/m^2 (inclusive)

Exclusion Criteria:

* Female subject who is pregnant, or plans to become pregnant during the study, or lactating, or sexually active with childbearing potential who is not using a medically accepted birth control method. Male subjects who are planning a partner pregnancy during the study
* Subjects receiving any live (includes attenuated) vaccination within the 8 weeks prior to Baseline (eg, inactivated influenza and pneumococcal vaccines are allowed but nasal influenza vaccination is not permitted). Live vaccines are not allowed during the study or for 20 weeks after the last dose of study drug
* Subject has received any investigational drug or experimental procedure within 90 days or 5 half-lives, whichever is longer, prior to IMP administration
* Subject has a known hypersensitivity to any components of the IMP as stated in this protocol
* Subject has a current or past history of gastrointestinal ulceration or other gastrointestinal disease
* Subject has cardiovascular or cerebrovascular disease, including hypertension, angina, ischemic heart disease, transient ischemic attacks, stroke, peripheral arterial disease sufficient to cause symptoms, and/or requires therapy to maintain stable status
* Subject has an active infection (eg, sepsis, pneumonia, abscess) or has had a serious infection (resulting in hospitalization or requiring parenteral antibiotic treatment) within 6 weeks prior to IMP administration
* Study participant has a history of a positive tuberculosis (TB) test or evidence of possible TB or latent TB infection at the Screening Visit
* Subject has concurrent acute or chronic viral hepatitis B or C or human immunodeficiency virus (HIV) infection
* Subject has 12-lead ECG with changes considered to be clinically significant at Screening Visit and Day -1
* Subject has active neoplastic disease or history of neoplastic disease within 5 years of Screening Visit (except for basal or squamous cell carcinoma of the skin or carcinoma in situ that has been definitively treated with standard of care)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2016-06-17 (Actual); Study Completion 2016-06-17 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events including injection site reactions and systemic injection reactions | From Screening Period (Day -21) until end of Safety-Follow-Up Visit (up to Day 85)
  An Adverse Event is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment.
Relative Bioavailability (BA) of Bimekizumab | Pre-dose (Day 1) until end of Safety-Follow-Up Visit (up to Day 85)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, Individual Patient Data cannot be adequately anonymized and there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.